CLINICAL TRIAL: NCT07064213
Title: Effect of an Informative Video About Perineal Tears on Anxiety During Labor: A Randomized Controlled Trial
Brief Title: An Informative Video About Perineal Tears During Labor for Anxiety Reduction: A Randomized Controlled Trial
Acronym: VITAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, ilia kleiner, Specialist Obstetrician & Gynecologist; Director, Labor and Delivery Rooms and Maternity Department, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WOMC-0109-25
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
Keywords: Perineal Tears; Childbirth Education; Primiparous Women; Labor and Delivery; Childbirth-Related Anxiety; Intrapartum Anxiety; Obstetric trauma; Episiotomy; Vaginal delivery; OASIS; STAI-S; Maternal mental health
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Participants watch an educational video about perineal tears and episiotomy via QR code before active labor.
  Interventions: Behavioral: Behavioral: Educational Video
- Control Group (No Intervention): Receives standard care without video

INTERVENTIONS:
Behavioral: Behavioral: Educational Video — Participants will watch a 2-minute educational video in Hebrew about perineal tears and episiotomy. The video includes information about types and grades of tears, risk factors, prevention strategies, episiotomy use, healing process, and when to seek help. The video is presented on a secure mobile device by the research team before the onset of active labor.
  Arms: Video Group

SUMMARY:
This study evaluates the impact of an informative video about perineal tears on maternal anxiety during labor. Perineal trauma during childbirth, especially severe tears such as obstetric anal sphincter injuries (OASIS), is associated with significant physical and psychological consequences, including anxiety, shame, fear, and social isolation. Despite growing awareness, many women report inadequate knowledge and preparation regarding these outcomes before labor.

This prospective, single-center, randomized controlled trial will be conducted at Edith Wolfson Medical Center in Holon, Israel. A total of 110 primiparous women admitted for induction or early labor will be recruited prior to the active phase of labor. Participants will be randomized into two groups in a 1:1 ratio. The intervention group will watch a 2-minute educational video explaining the types, implications, and prevention strategies related to perineal tears. The control group will receive standard care without video exposure.

The primary objective is to assess change in maternal anxiety using the validated State-Trait Anxiety Inventory (STAI-S) questionnaire, measured at baseline and 2-24 hours postpartum. Secondary outcomes include satisfaction with the video (in the intervention group), rates of perineal tears, episiotomy, and OASIS. Data will be collected from the hospital's EMR system and patient-reported questionnaires, stored securely and coded. The study aims to determine whether increasing knowledge through a short educational intervention can reduce childbirth-related anxiety and improve the birth experience.

DETAILED DESCRIPTION:
Background and Rationale:

Perineal tears during vaginal delivery are a common obstetric complication, affecting both the physical and emotional well-being of mothers. Numerous studies have highlighted the psychological burden associated with severe tears, including obstetric anal sphincter injuries (OASIS). These can result in postpartum depression, posttraumatic stress symptoms (PTS), anxiety, and disruption to intimate and social relationships.

A comprehensive review by Darmody et al. (2020) and qualitative synthesis by Priddis et al. (2013) have shown that women experiencing significant perineal trauma may report feelings of shame, loneliness, failure, and fear, often amplified by insufficient understanding or preparation before delivery. More recent studies (Opondo et al., 2023; Baumann et al., 2024) found that the severity of tears correlates with psychological morbidity postpartum, including childbirth-related PTSD.

These findings underscore the importance of providing accessible, accurate information to women before delivery to empower them, reduce fear, and foster realistic expectations. However, no randomized controlled trial has yet evaluated whether a brief, targeted educational intervention specifically about perineal tears can reduce anxiety when given just before the active phase of labor.

Study Objective:

To evaluate whether viewing a short, informative video about perineal tears before the onset of active labor reduces maternal anxiety.

Study Design:

This is a prospective, randomized controlled trial (RCT) with two parallel arms. The study will be conducted at Edith Wolfson Medical Center, Holon, Israel, over a 12-month period. A total of 110 primiparous women ≥18 years old at ≥37 weeks gestation will be recruited from the Maternal-Fetal Medicine Unit or Delivery Room prior to active labor.

Eligibility Criteria:

Inclusion:

Primiparous women

Age 18-45

Gestational age ≥37 weeks

Fluent in Hebrew (able to complete STAI-S questionnaire)

Exclusion:

Intrauterine fetal death

Termination of pregnancy

Known anxiety disorder

Language barrier

Cesarean section during labor

Withdrawal of consent

Randomization:

Participants will be randomly assigned (1:1) to the intervention or control group. Randomization will be done using computerized block randomization by the study team.

Intervention:

The intervention group will watch a 2-minute educational video (in Hebrew) produced by the research team. The video provides information on types and degrees of perineal tears, the role of episiotomy, possible symptoms, healing, and preventative techniques. Viewing will take place using the researchers' secure mobile device.

The control group will receive routine intrapartum care with no additional information.

Outcomes:

Primary Outcome:

Change in STAI-S anxiety score from before active labor to 2-24 hours postpartum

Secondary Outcomes:

Satisfaction with the video (intervention group only)

Rate of perineal tears (any grade)

Rate of episiotomy

Rate of obstetric anal sphincter injuries (OASIS)

Data Collection and Analysis:

Anxiety will be assessed using the validated Hebrew version of the STAI-S questionnaire at two time points:

At enrollment, before active labor

2-24 hours after delivery

Demographic, clinical, and birth data will be extracted from the Chameleon hospital EMR system. Data will include: age, BMI, parity, pregnancy complications, labor duration, birthweight, Apgar scores, pH umbilical, and neonatal unit admission. All data will be anonymized and stored on password-protected hospital systems.

Statistical analysis will use SPSS v30. Continuous variables will be compared using t-tests, categorical variables with chi-square tests. p < 0.05 will be considered statistically significant.

Sample Size Justification:

A pilot evaluation of 10 women showed mean STAI-S scores of 41 (SD = 11). Assuming a 15% reduction in anxiety in the intervention group, with α=0.05 and 80% power, 100 participants are required. Accounting for 10% loss to follow-up, the final sample is 110 (55 per arm).

Ethics and Privacy:

All participants will provide informed consent before enrollment. Data will be stored in coded form, with no personal identifiers. Participants may withdraw at any point. Ethics approval is/will be granted by the Wolfson Medical Center Helsinki Committee.

The study is expected to contribute valuable data on whether a low-cost, scalable educational tool can reduce childbirth anxiety and improve maternal emotional outcomes.

ELIGIBILITY:
Inclusion:

Primiparous women

Age ≥18

Gestational age ≥37 weeks

Fluent in Hebrew (able to complete STAI-S)

Exclusion:

IUFD

Pregnancy termination

Diagnosis of anxiety disorder

Language barrier (cannot complete STAI-S)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified women who are pregnant and meet inclusion criteria for labor participation.
Enrollment: 110 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Change in maternal anxiety score | 2-24 hours postpartum
  The primary outcome is the change in maternal anxiety as measured by the State-Trait Anxiety Inventory - State version (STAI-S). This validated questionnaire includes 20 items that assess situational anxiety on a 4-point scale, with total scores ranging from 20 to 80. Higher scores indicate greater anxiety. The STAI-S will be administered at two time points: (1) upon enrollment, before the active phase of labor begins, and (2) 2 to 24 hours after delivery. The difference in scores between these two time points will be compared between the intervention and control groups to assess whether viewing a short, informative video about perineal tears reduces anxiety during labor.

SECONDARY OUTCOMES:
Satisfaction with video (intervention group only) | 2-24 hours postpartum
  Satisfaction with the educational video will be assessed in the intervention group only. Participants will complete a brief, structured questionnaire within 2 to 24 hours postpartum. The questionnaire includes items assessing perceived usefulness, clarity of information, emotional impact, and whether the video helped them feel more prepared for labor and perineal outcomes.
Rate of perineal tears | During delivery
Rate of episiotomy | During delivery
Rate of OASIS | During delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Kleiner, MD, Principal Investigator — Wolfson Medical Center; Hagit Eisenberg, MD, Study Director — Wolfson Medical Center; Julia Barda Fishler, MD, Study Director — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include STAI-S questionnaire scores at both time points, participant age, gestational age at delivery, mode of delivery, and perineal outcomes including episiotomy, perineal tear grade, and OASIS status. No personally identifiable information will be shared. Data will be available upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after study completion and available for 2 years.
Access Criteria: De-identified individual participant data and supporting documents (study protocol, SAP, and informed consent form) will be made available to qualified researchers with institutional ethics approval. Access will be granted upon submission and approval of a methodologically sound proposal. Requests should be sent to the principal investigator via email. Approved data will be shared electronically in a secure, password-protected format.

REFERENCES:
- [Background] Opondo C, Harrison S, Sanders J, Quigley MA, Alderdice F. The relationship between perineal trauma and postpartum psychological outcomes: a secondary analysis of a population-based survey. BMC Pregnancy Childbirth. 2023 Sep 6;23(1):639. doi: 10.1186/s12884-023-05950-6. PMID 37674105
- [Background] Priddis H, Dahlen H, Schmied V. Women's experiences following severe perineal trauma: a meta-ethnographic synthesis. J Adv Nurs. 2013 Apr;69(4):748-59. doi: 10.1111/jan.12005. Epub 2012 Oct 12. PMID 23057716
- [Background] Darmody E, Bradshaw C, Atkinson S Dr. Women's experience of obstetric anal sphincter injury following childbirth: An integrated review. Midwifery. 2020 Dec;91:102820. doi: 10.1016/j.midw.2020.102820. Epub 2020 Aug 22. PMID 32861872